CLINICAL TRIAL: NCT03105440
Title: Innovation Oncological Rehabilitation: Applicability of the Different Techniques Physiotherapeutic Post Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 41887715.0.0000.5503
Record Dates: First submitted 2016-06-01; First posted 2017-04-10 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Lymphedema; Pain
Keywords: breast cancer; lymphedema; pain; range of motion; technologic innovation; rehabilitation
MeSH Terms: conditions — Lymphedema; Pain; Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Robotic rehabilitation (Experimental): It Will be used a exoskeleton Armeo®Spring, to training to affected upper limb, the protocol of the treatment is constituted for 8 games. The equipment arm will be adjusted the volunteers height, in sitting position, allowing support against the action of gravity of the arm and forearm, supporting 45° of the shoulder flexion, which will be facilitation the member movement.
  Interventions: Other: Robotic rehabilitation
- Virtual reality (Experimental): The software used in this study was developed by the members of the Laboratory of Sensory and Motor Engineering Rehabilitation Together with Federal University of Uberlândia. This virtual reality of projection software, which uses Kinact®, captures the patient's picture and transfers to the monitor. The exercises provided by game are similar to those performed in conventional therapy; however, in a more entertaining form.
  Comprised 8 exercises to upper limbs and trunk. The patient should reach the red circle until it becomes green.
  Interventions: Other: Virtual reality
- Vibration therapy (Experimental): The vibration mat used in this study was developed by the members of the Laboratory of Sensory and Motor Engineering Rehabilitation together with mark Vibra Ind. e Com. Prod. Electronics Ltda.
  Will participate 20 woman, that stay in supine position, with the enveloped member of the vibration mat, elevated and supported. The volunteer will be submitted to 15 minutes of vibration with frequency of the 40 hertz, in both upper limbs.
  Interventions: Other: Vibration therapy
- Hand cycling (Experimental): Will participate 20 woman, submitted hand cycling through of the adapted bicycle to upper members. The protocol will be comprised by track without obstacle, comprised by 10 turns. The cyclic movement velocity will be realized according to the physical fatigue of patients.
  Interventions: Other: Hand cycling
- Control group (Experimental): Will participate 20 healthy woman, that won't pass to the treatment physiotherapeutic, only will be collected the electromyography and dynamometer.
  Interventions: Other: Control group
- Canoeing (Experimental): Will participate 20 woman, submitted canoeing activates, through rowing realized in therapeutic pool, with the aid and supervision of the therapeutic. It is important highlight that the exercises intensity will be to realized according to the physical fatigue of patients.
  Interventions: Other: Canoeing

INTERVENTIONS:
Other: Virtual reality — This virtual reality of projection software, which uses Kinact®, captures the patient's picture and transfers to the monitor. The exercises provided by game are similar to those performed in conventional therapy; however, in a more entertaining form.
  Comprised 8 exercises to upper limbs and trunk. The patient should reach the red circle until it becomes green.
  Arms: Virtual reality
Other: Vibration therapy — The vibration mat used in this study was developed by the members of the Laboratory of Sensory and Motor Engineering Rehabilitation together with mark Vibra Ind. e Com. Prod. Electronics Ltda.
  Will participate 20 woman, that stay in supine position, with the enveloped member of the vibration mat, elevated and supported. The volunteer will be submitted to 15 minutes of vibration with frequency of the 40 hertz, in both upper limbs.
  Arms: Vibration therapy
Other: Hand cycling — Will participate 20 woman, submitted hand cycling through of the adapted bicycle to upper members. The protocol will be comprised by track without obstacle, comprised by 10 turns. The cyclic movement velocity will be realized according to the physical fatigue of patients.
  Arms: Hand cycling
Other: Canoeing — Will participate 20 woman, submitted canoeing activates, through rowing realized in therapeutic pool, with the aid and supervision of the therapeutic. It is important highlight that the exercises intensity will be to realized according to the physical fatigue of patients.
  Arms: Canoeing
Other: Robotic rehabilitation — It Will be used a exoskeleton Armeo®Spring, to training to affected upper limb, the protocol of the treatment is constituted for 8 games. The equipment arm will be adjusted the volunteers height, in sitting position, allowing support against the action of gravity of the arm and forearm, supporting 45° of the shoulder flexion, which will be facilitation the member movement.
  Arms: Robotic rehabilitation
Other: Control group — Will participate 20 healthy woman, that won't pass to the treatment physiotherapeutic, only will be collected the electromyography and dynamometer.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effects and validate news physiotherapy techniques: robotic rehabilitation, virtual reality, vibration therapy, canoeing and hand cycling in the secondary clinical complications of the breast cancer, through the Biomedical Instrumentation. It will be realized the double-blind longitudinal clinical study. Will participate in the study 100 women post breast cancer surgery, the volunteers will be allocated in the respective modalities treatment; and 20 healthy volunteers, will be only the control group. The volunteers conducted 10 physiotherapy session, and it will be evaluated after, during and before of the treatment, to evaluated myoelectric activity, scapular and hand muscle strength, range of motion, circumference of the upper limbs and quality of life. Expected to Positive Results With regard to the minimization of pain intensity and lymphedema, favoring the improvement of range of motion of the shoulder joint, myoelectric activity, increased muscle strength, and consequently improves the quality of life.

DETAILED DESCRIPTION:
The brest cancer is considered a public health problem worldwide. In Brazil, there was increased survival due to advances in early diagnosis and the therapeutic approaches each more accurate and effective, however these women require care and attention for short and long time, due to the consequences physical and psychosocial, que undertake their quality of life. The innovative techniques physiotherapy treatment can contribute to the prevention and treatment of complications, with the intention to facilitate the early return of women to their daily activities. The aim of this study is to evaluate the effects and validate news physiotherapy techniques: robotic rehabilitation, virtual reality, vibration therapy, canoeing and hand cycling in the secondary clinical complications of the breast cancer, through the Biomedical Instrumentation. It will be realized the double-blind longitudinal clinical study. Will participate in the study 100 women post breast cancer surgery, the volunteers will be allocated in the respective modalities treatment; and 20 healthy volunteers, will be only the control group. The volunteers conducted 10 physiotherapy session, and it will be evaluated after, during and before of the treatment, to evaluated myoelectric activity, scapular and hand muscle strength, range of motion, circumference of the upper limbs and quality of life. Expected to Positive Results With regard to the minimization of pain intensity and lymphedema, favoring the improvement of range of motion of the shoulder joint, myoelectric activity, increased muscle strength, and consequently improves the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Conservative or non-conservative breast cancer surgery;
* Acceptance of the Informed Consent.

Exclusion Criteria:

* Patients who still have chest drain;
* Volunteers who need any aiding device to remain in orthostatism;
* Patients don't accepted of the Informed Consent;
* Patients who ar afraid of water.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-04 (Actual); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Edema | 10th. day.
  Was measure thought perimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Izabela S. Mendes, Study Director — Universidade do Vale do Paraíba
Locations (1):
- University of Vale do Paraíba, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No